CLINICAL TRIAL: NCT04554979
Title: Corona Virus (COVID-19) Disease Duration and Gastrointestinal Tract (GIT) Manifestations; Can be New Disease Severity Classification. A Pilot Egyptian Single National Center Experience
Brief Title: COVID-19 Disease Duration and GIT Manifestations. A New Disease Severity Classification. An Egyptian Experience
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Hegazy, Professor of Internal Medicine Hepatology & gastroenterology Unit Faculty of medicine, Cairo University
Other Study IDs: 1004
Record Dates: First submitted 2020-09-12; First posted 2020-09-18 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Covid19; Diarrhea
Keywords: COVID-19 disease outcomes and duration; GIT manifestations; Diarrhea
MeSH Terms: conditions — COVID-19; Diarrhea | interventions — Hydroxychloroquine; Adrenal Cortex Hormones; Anticoagulants; Anti-Bacterial Agents; Ascorbic Acid; Zinc

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Duration of COVID-19 symptoms less than 12 days
  Interventions: Drug: Hydroxychloroquine Pill
- Group 2: Duration of COVID-19 symptoms equal or more than 12 days
  Interventions: Drug: Hydroxychloroquine Pill

INTERVENTIONS:
Drug: Hydroxychloroquine Pill — hydroxychloroquine 400 mg twice daily first day and maintained on 200 mg twice daily for 6 days in mild cases and 10 days in moderate cases. Also they received anticoagulants, vitamin c and zinc. In case of secondary bacterial infection, empiric antibiotics are started
  Other Names: corticosteroids; anticoagulant; antibiotic; vitamin c pill; zinc pill

SUMMARY:
The present study conducted to correlate symptoms not only constitutional and respiratory, but GIT as a principle presentation, with laboratory markers and COVID-19 severe acute respiratory syndrome (SARS-COV2) disease outcomes, as the duration of symptoms varies substantially between patients; the investigators undertook this study to determine the optimal time to predict COVID-19 outcomes based on real-time experience.

DETAILED DESCRIPTION:
This observational retrospective cohort single center national study was conducted on patients who tested positive COVID-19 infection by the polymerase chain reaction (PCR) of nasopharyngeal sample in the period from first June to the med of July 2020. Patients were recruited from Kasr Al-Aini School of medicine, COVID-19 out-patient clinic, Cairo University hospitals.

The diagnosis and classification of severity of COVID-19 infection were made according to the clinical management of COVID-19, released by the World Health Organization (WHO), mild and moderate case were recruited, the treatment protocol used was according to the Egyptian ministry of health treatment recommendations, which met in part the criteria that was later on published by the national institute of health, Mild and moderate cases once diagnosed by PCR received hydroxychloroquine 400 mg twice daily first day and maintained on 200 mg twice daily for 6 days in mild cases and 10 days in moderate cases. Also they received anticoagulants, vitamin c and zinc. In case of secondary bacterial infection, empiric antibiotics are started till result of sputum culture and sensitivity. Steroids were initiated in hypoxic cases that required supplemental oxygen and in cases of persistent symptoms.

Any adult patient (age ≥18 years) suffering from mild or moderate COVID-19 infection was included in this study. While severe cases according to WHO classifications and patients aged less than18 were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Mild and moderate COVID-19 patients:

Exclusion Criteria:

* Age less than 18 years
* Severe COVID-19 patients: with dyspnea, hypoxia, or >50 percent lung involvement on imaging within 24 to 48 hours
* Critical COVID-19 patients: with respiratory failure, shock, or multiorgan dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients was recruited from COVID19 out-patient clinic, Cairo University hospitals. Severity Classification made according to the WHO (13) and Egyptian ministry of health treatment recommendations (14) Clinical data was collected including patient demographics (age, gender, weight and height, body mass index, comorbid conditions (e.g.diabetes mellitus, chronic pulmonary disease), vital signs. Clinical symptoms were recorded using yes/no checklist about constitutional symptoms, respiratory symptoms, loss of taste, loss of smell and gastrointestinal symptoms.The patients were followed up daily; by telehealth through phone calls and commercial video chat platforms, till symptoms offset. Laboratory assessment was collected within 24 hours of symptoms onset (complete blood picture, kidney and liver biochemistry, random blood sugar, serum C-reactive protein, D-dimer, ferritin, lipid profile, and lactate dehydrogenase). CT chest was performed and its result was recorded
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
COVID-19 disease spectrum and duration | july 2020 to june 2020
  The investigators tried to correlate disease severity with disease duration
GIT manifestations among COVID-19 patients | july 2020 to june 2020
  spectrum of GIT manifestations in COVID-19 patients was investigated

SECONDARY OUTCOMES:
Non-communicable disease and COVID-19 | july 2020 to june 2020
  The link between non-communicable disease (including diabetes, hypertension and Hypercholesterolemia) severity and COVID-19 prognosis
Seasonal change and COVID-19 | july 2020 to june 2020
  the investigators studied the Impact of weather climate on COVID-19 presentations (higher incidence of diarrhea in COVID-19 patients in summer) and outcomes
Possible region specific classification for COVID-19 disease | july 2020 to june 2020
  The investigators tried to find new Egyptian classification fro COVID-19 disease severity

CONTACTS AND LOCATIONS:
Overall Officials: Mona M Hegazy, MD, Principal Investigator — Professor of Internal Medicine Hepatology & gastroenterology Unit. Faculty of medicine Cairo University; Ahmed M Abdul Ghani, MD, Study Director — Lecturer of Internal Medicine Hepatology & gastroenterology Unit. Faculty of medicine Cairo University; Rania M Lithy, MD, Study Chair — Lecturer of Endemic medicine and hepatogastroenterology. Faculty of medicine Cairo University; Hoda M abdel-Hamid, MD, Study Chair — Lecturer of Respiratory medicine. Faculty of medicine Cairo University; Mahmoud Wahba, MD, Study Chair — Lecturer of Internal Medicine Division of Gastroenterology, Kasr Alainy . Faculty of Medicine, Cairo University; Omar Ashoush, MD, Study Chair — Lecturer of Internal Medicine Hepatology & gastroenterology Unit. Faculty of medicine Cairo University; Mohamed Tharwat Hegazy, MD, Study Chair — Lecturer of Internal Medicine Department, Rheumatology and Clinical Immunology unit, Faculty of Medicine, Cairo University
Locations (1):
- Faculty of Medicine Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1.World Health Organization. Novel coronavirus (2019-nCoV): situation report-40. Available at: https://www.who.int/docs/default-source/coronaviruse/situation-reports/20200229-sitrep-40-covid-19.pdf. Accessed 29 February 2020.
- [Background] Hoehl S, Rabenau H, Berger A, Kortenbusch M, Cinatl J, Bojkova D, Behrens P, Boddinghaus B, Gotsch U, Naujoks F, Neumann P, Schork J, Tiarks-Jungk P, Walczok A, Eickmann M, Vehreschild MJGT, Kann G, Wolf T, Gottschalk R, Ciesek S. Evidence of SARS-CoV-2 Infection in Returning Travelers from Wuhan, China. N Engl J Med. 2020 Mar 26;382(13):1278-1280. doi: 10.1056/NEJMc2001899. Epub 2020 Feb 18. No abstract available. PMID 32069388
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Shi H, Han X, Jiang N, Cao Y, Alwalid O, Gu J, Fan Y, Zheng C. Radiological findings from 81 patients with COVID-19 pneumonia in Wuhan, China: a descriptive study. Lancet Infect Dis. 2020 Apr;20(4):425-434. doi: 10.1016/S1473-3099(20)30086-4. Epub 2020 Feb 24. PMID 32105637
- [Background] Jin X, Lian JS, Hu JH, Gao J, Zheng L, Zhang YM, Hao SR, Jia HY, Cai H, Zhang XL, Yu GD, Xu KJ, Wang XY, Gu JQ, Zhang SY, Ye CY, Jin CL, Lu YF, Yu X, Yu XP, Huang JR, Xu KL, Ni Q, Yu CB, Zhu B, Li YT, Liu J, Zhao H, Zhang X, Yu L, Guo YZ, Su JW, Tao JJ, Lang GJ, Wu XX, Wu WR, Qv TT, Xiang DR, Yi P, Shi D, Chen Y, Ren Y, Qiu YQ, Li LJ, Sheng J, Yang Y. Epidemiological, clinical and virological characteristics of 74 cases of coronavirus-infected disease 2019 (COVID-19) with gastrointestinal symptoms. Gut. 2020 Jun;69(6):1002-1009. doi: 10.1136/gutjnl-2020-320926. Epub 2020 Mar 24. PMID 32213556
- [Background] Pan L, Mu M, Yang P, Sun Y, Wang R, Yan J, Li P, Hu B, Wang J, Hu C, Jin Y, Niu X, Ping R, Du Y, Li T, Xu G, Hu Q, Tu L. Clinical Characteristics of COVID-19 Patients With Digestive Symptoms in Hubei, China: A Descriptive, Cross-Sectional, Multicenter Study. Am J Gastroenterol. 2020 May;115(5):766-773. doi: 10.14309/ajg.0000000000000620. PMID 32287140
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] 9. Mo P, Xing Y, Xiao Y, et al. Clinical characteristics of refractory COVID-19 pneumonia in Wuhan, China. [published online ahead of print, 2020 Mar 16]. Clin Infect Dis 2020:ciaa270. doi:10.1093/ 54. cid/ciaa270
- [Background] D'Amico F, Baumgart DC, Danese S, Peyrin-Biroulet L. Diarrhea During COVID-19 Infection: Pathogenesis, Epidemiology, Prevention, and Management. Clin Gastroenterol Hepatol. 2020 Jul;18(8):1663-1672. doi: 10.1016/j.cgh.2020.04.001. Epub 2020 Apr 8. PMID 32278065
- [Background] Tian S, Chang Z, Wang Y, Wu M, Zhang W, Zhou G, Zou X, Tian H, Xiao T, Xing J, Chen J, Han J, Ning K, Wu T. Clinical Characteristics and Reasons for Differences in Duration From Symptom Onset to Release From Quarantine Among Patients With COVID-19 in Liaocheng, China. Front Med (Lausanne). 2020 May 12;7:210. doi: 10.3389/fmed.2020.00210. eCollection 2020. PMID 32574322
- [Background] Lu Y, Li Y, Deng W, Liu M, He Y, Huang L, Lv M, Li J, Du H. Symptomatic Infection is Associated with Prolonged Duration of Viral Shedding in Mild Coronavirus Disease 2019: A Retrospective Study of 110 Children in Wuhan. Pediatr Infect Dis J. 2020 Jul;39(7):e95-e99. doi: 10.1097/INF.0000000000002729. PMID 32379191
- [Background] 13. World Health Organization. Clinical management of COVID-19: interim guidance. 2020, p.62.
- [Background] Coronavirus Disease 2019 (COVID-19) Treatment Guidelines [Internet]. Bethesda (MD): National Institutes of Health (US); 2021 Apr 21-2024 Mar 1. Available from http://www.ncbi.nlm.nih.gov/books/NBK570371/ PMID 34003615
- [Background] World Medical Association Inc. Declaration of Helsinki. Ethical principles for medical research involving human subjects. J Indian Med Assoc. 2009 Jun;107(6):403-5. No abstract available. PMID 19886379